CLINICAL TRIAL: NCT00261521
Title: Double-blind Study to Assess the Impact of Normalization of Hemoglobin Compared to Partial Correction of Hemoglobin With EPREX�/ERYPO� on Left Ventricular Structure in Early Hemodialysis Patients (RWJ-22512)
Brief Title: A Study of the Safety and Efficacy of Long-term Correction of Anemia With Epoetin Alfa in Early Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004420
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Kidney Failure, Chronic; Anemia
Keywords: Kidney failure, Chronic; End-stage renal disease; Kidney failure; Anemia; Dialysis; Epoetin; Erythropoetin; Epoetin alfa
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia; Renal Insufficiency | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study in early hemodialysis patients (on dialysis 3 to 18 months) is to assess the effect of correction versus partial correction of anemia using epoetin alfa on heart pumping function.

DETAILED DESCRIPTION:
Cardiovascular disease is very common among patients with end-stage renal disease. This study is a long-term, double-blind, parallel-group, multicenter study to determine the efficacy and safety of administering epoetin alfa to treat anemia (patients in Group 1) or partially treat anemia (patients in Group 2) in order to reduce the risk of heart failure in chronic renal failure patients on early dialysis and to improve their quality of life. Efficacy of epoetin alfa will be determined by comparing between Group 1 and Group 2 the heart structure (changes in left ventricle volume and mass viewed on echocardiograms), development of heart failure, correlation between changes in heart structure and hemoglobin level, a 6-minute walking test, and by 2 quality of life measures-a quality of life questionnaire and a fatigue questionnaire. Safety data associated with elevation of hemoglobin will be collected and monitored throughout the study: hemoglobin-related adverse events include thrombovascular events, seizures, and hypertension. Development of antibodies to erythropoetin over long-term treatment also will be assessed by serum samples gathered over the course of the study. The hypothesis of this study is that earlier and longer-term anemia intervention in patients without symptomatic heart disease or heart architecture distortions may conserve heart function and improve their quality of life, and that the intervention will be well tolerated by the patients. Patients not on epoetin alfa at start: epoetin alfa (50 IU/kg), 3 times per week with increases every 4 weeks at either 25 IU/kg or up to 25% of previous dose to reach target hemoglobin (Hb), then dose maintained. Patients on or switched to epoetin alfa at start are titrated to maintain target Hb.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis for 3 to 18 months and expected to remain on hemodialysis for at least two more years and with a life expectancy of a year or more
* Kidney transplant patients, whose transplant has failed, and now have been on hemodialysis for 3-18 months, may be eligible for the study, if they are not receiving excessive immunosuppression (e.g., <=10 mg of steroids/day allowed)
* Pre-dialysis hemoglobin 8-12 g/dL, inclusive, within the previous month (single reading is sufficient)
* Stable hemodialysis vascular access, within the previous 3 months
* No heart disease or asymptomatic heart disease without enlarged heart

Exclusion Criteria:

* Heart diseases for which surgical intervention occurred during the previous two years or which may require intervention within the next year
* Patients with medical conditions likely to affect the response to epoetin
* Predialysis sitting diastolic blood pressure >= 100 mmHg on average for the previous month
* Folate, Vitamin B12, or transferrin deficiency
* History of seizure within 1 year
* Transfusion within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2000-02; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Percent change in left ventricular volume index (LVVI) at Week 96.

SECONDARY OUTCOMES:
Percent change at Week 96 in left ventricular mass index (LVMI), development of new heart failure, correlation between change in left ventricular indices and average maintenance hemoglobin, 6-minute walking test, and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Parfrey PS, Foley RN, Wittreich BH, Sullivan DJ, Zagari MJ, Frei D. Double-blind comparison of full and partial anemia correction in incident hemodialysis patients without symptomatic heart disease. J Am Soc Nephrol. 2005 Jul;16(7):2180-9. doi: 10.1681/ASN.2004121039. Epub 2005 May 18. PMID 15901766
- [Derived] Williams CE, Curtis BM, Randell EW, Foley RN, Parfrey PS. Cardiac biomarkers and health-related quality of life in new hemodialysis patients without symptomatic cardiac disease. Can J Kidney Health Dis. 2014 Jul 15;1:16. doi: 10.1186/2054-3581-1-16. eCollection 2014. PMID 26038709